CLINICAL TRIAL: NCT05546372
Title: Endobiliary Radiofrequency Ablation for Malignant Biliary Obstruction Due to Perihilar Cholangiocarcinoma: a Randomized Controlled Trial
Brief Title: Endobiliary Radiofrequency Ablation for Malignant Biliary Obstruction Due to Perihilar Cholangiocarcinoma
Acronym: RACCOON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Rogier P. Voermans, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL76591.029.22
Record Dates: First submitted 2022-08-25; First posted 2022-09-19 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Perihilar Cholangiocarcinoma
Keywords: Endobiliary radiofrequency ablation; Stent patency
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endobiliary RFA + stent placement (Experimental)
  Interventions: Device: Endobiliary radiofrequency ablation (eRFA); Device: uncovered self-expanding metal stent (uSEMS)
- Stent placement only (Active Comparator)
  Interventions: Device: uncovered self-expanding metal stent (uSEMS)

INTERVENTIONS:
Device: Endobiliary radiofrequency ablation (eRFA) — Intraductal radiofrequency ablation of tumor prior to stent placement
  Arms: Endobiliary RFA + stent placement
Device: uncovered self-expanding metal stent (uSEMS) — Intraductal placement of uncovered metal stent

SUMMARY:
A multicentre, parallel group, open label, randomized controlled trial comparing endobiliary RFA prior to metal stent placement with stent placement only in patients with inoperable perihilar cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Capable of providing written and oral informed consent.
* Histological or cytological proof of perihilar CCA (adenocarcinoma).
* Perihilar biliary obstruction with an indication for drainage with uSEMS.*
* Advanced (no candidate for surgical resection) due to metastases, vascular or lymph node (N2) involvement on imaging or during staging laparoscopy according to multidisciplinary team (MDT).

  * Only patients with pCCA are eligible however in case of reasonable doubt between intrahepatic CCA with a perihilar biliary obstruction or massforming pCCA, patients can be included.

Exclusion Criteria:

* Patients who potentially qualify for curative resection of pCCA.
* pCCA eligible for liver transplantation.
* Life-expectancy less than 3 months.
* ERCP and PTC technically not feasible.
* Uncontrolled coagulopathy (PTT >1,5x prolonged or thrombocytes below 40*10E9/L).
* Ongoing cholangitis or liver abscess. Patients are required to be off antibiotic treatment for cholangitis and/or liver abscess at least 7 days.
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study.
* Patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-11-09 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to biliary obstruction | Through study completion, max 1 year
  Defined as period between initial procedure and recurrence of biliary obstruction. Recurrence of biliary obstruction is defined as recurrent jaundice (conjugated bilirubin ≥ 40 umol/l (≥2.3 mg/dl)), presence of biochemical evidence of cholestasis along with dilatation of the drained bile duct(s), or endoscopic findings suggesting stent occlusion.

SECONDARY OUTCOMES:
Quality of life expressed in quality adjusted life-years (QALYs) | Through study completion, max 1 year
  EORTC QLQ-C30, BIL21 and EQ-5D questionnaires are to be filled out 4 weeks and every3 months after the intervention
Number of patients with technical success of initial ablation | During intervention
  Defined as completion of ablation of the malignant stenosis through which the stent will be placed using RFA for 120 seconds with 7W.
Number of patients with functional success | 14 days
  In case of inadequate drainage prior to the procedure (bilirubin ≥40 umol/L [≥2.3 mg/dl]), defined as 50% decrease or normalization of bilirubin level within 14 days of the procedure or relieve of symptoms in case of cholangitis. In case of sufficient drainage prior to the procedure, a persistent bilirubin level <40 umol/L (<2.3 mg/dl) after 14 days is considered functional success.
Presumed reason of recurrent biliary obstruction | Through study completion, an average of 1 year
  1. Stent occlusion due to tumour ingrowth
  2. Stent occlusion due to tumour overgrowth
  3. Stent occlusion due to sludge with/or without stones, hemobilia, food impaction
  4. Stent migration
Need for unscheduled re-intervention (PTC and/or ERCP) to achieve adequate biliary drainage. | Through study completion, an average of 1 year
Need for external drainage catheters. | Through study completion, an average of 1 year
Time to re-intervention. | Through study completion, an average of 1 year
Stent patency after repeated eRFA. | Through study completion, an average of 1 year
Adverse events within 30 days after the procedu | 30 days
Overall survival. | Through study completion
Healthcare costs. | Through study completion, max 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided